CLINICAL TRIAL: NCT06716775
Title: Tumor Treating Fields (TTF) in Combination with Stereotactic Radiosurgery(SRS) for Brain Metastases from Non-small Cell Lung Cancer: a Randomized, Controlled, Open-label Study.
Brief Title: Tumor Treating Fields (TTF) in Combination with Stereotactic Radiosurgery(SRS) for Brain Metastases from Non-small Cell Lung Cancer.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Healthy Life Innovation Medical Technology Co., Ltd (Industry)
Collaborators: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL-10
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: NSCLC Brain Metastasis
Keywords: TTF; NSCLC brain metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TTF+Best Standard of Care (Experimental)
  Interventions: Device: Tumor treating felds (TTF); Other: Best Standard of Care
- Best Standard of Care (Active Comparator)
  Interventions: Other: Best Standard of Care

INTERVENTIONS:
Device: Tumor treating felds (TTF) — Tumor Treating Fields will be administered continuously with a planned ≥ 18 h per day.
  Arms: TTF+Best Standard of Care
Other: Best Standard of Care — Patients will be treated with the best known standard of care for NSCLC brain metastasis and undergo SRS alone.

SUMMARY:
This is a randomized, controlled, open-label, phase III trials. The main purpose of this study is to evaluate the effectiveness and safety of tumor treating felds (TTF) combined with stereotactic radiosurgery (SRS) in the treatment of brain metastases from non-small cell lung cancer (NSCLC) .

ELIGIBILITY:
Inclusion Criteria:

1. The age of the subject was between 18 and 75 years old (inclusive), regardless of gender;
2. The predicted survival time was ≥3 months;
3. Newly diagnosed with NSCLC brain metastasis;
4. MRI imaging showed 1-10 unresectable brain metastases;
5. Karnofsky performance status (KPS) score ≥70;
6. Able to operate the TTF independently or with the help of a caregiver;
7. Subjects of childbearing potential had to agree to use effective contraception for the duration of the trial;
8. Voluntarily signed the informed consent form.

Exclusion Criteria:

1. Positive driver genes;
2. Recurrent brain metastasis of NSCLC;
3. Suffering from severe cerebral edema;
4. Leptomeningeal metastases;
5. Participants had to meet certain criteria for bone marrow, liver and kidney function before enrollment, and were not eligible if they had any of the following:

   1. platelet count < 100×103/μL;
   2. absolute neutrophil count < 1.5×103/μL;

   d. AST or ALT exceeding 2.5 times the upper limit of normal; c.Total bilirubin more than 1.5 times the upper limit of the normal range; d.Severe renal impairment (serum creatinine >1.7 mg/dL, or >150 μmol/L);
6. There were infection, ulcer and unhealed wound in the skin where the electrode was applied；
7. Patients allergic to conductive hydrogels or medical adhesives;
8. Those who are pregnant or preparing to become pregnant or who are breastfeeding;
9. Patients with poor compliance, as judged by the investigator, or other factors considered by the investigator to be not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Intracranial tumor progression-free survival (iPFS) | 3 years
  Defined as the time from randomization to the first occurrence of intracranial progression (according to RANO-BM criteria) or neurologic death, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  Defined as the time from the date of treatment until death due to any cause.
Objective response rate (ORR) | 3 years
  Defined as the number (%) of patients with at least 1 visit response of complete response (CR) or partial response (PR).
Time to neurocognitive failure | 3 years
Rate of intracranial progression at 2, 4, 6, 8, 10, 12 months | 3 years
Neurocognitive failure-free survival | 3 years
Rate of decline in cognitive function | 3 years
Number of participants with adverse events (AEs) | 3 years
  Adverse events will be defined as the incidence, frequency and severity of adverse events (AEs) noted in patients treated with study treatments

IPD SHARING:
Plan to Share IPD: Undecided